CLINICAL TRIAL: NCT04085640
Title: Obturator Nerve Block in Total Hip Arthrosplasty. a Randomized Controlled Double Blind Study
Brief Title: Obturator Nerve Block in Total Hip Arthrosplasty
Acronym: NOCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Medipole Garonne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NOCH
Record Dates: First submitted 2019-09-03; First posted 2019-09-11 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Primary Total Hip Arthroplasty
Keywords: Hip Arthroplasty; regional anesthesia; obturator nerve block
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obturator nerve block with Ropivacaine (Experimental): Obturator nerve block will be performed before general anesthesia as descripted by Nielsen (RAPM, 2019). A linear transducer will be oriented in the transverse plane and placed in the inguinal crease. The tail of the transducer will be tilted distal in order to visualize the pectineus muscle (medial to the femoral vessels) at its insertion at the superior pubic ramus superficial to the external obturator muscle. An 80 mm nerve block needlewill be inserted in-plane from the lateral end of the transducer and advanced until the tip of the needle will be inside the interfascial plane between the pectineus and the obturator externus muscles. 20 milliliters of ropivacaine 2 mg/mL will be injected in the interfacial plane between the pectineus and external obturator muscles.
  Interventions: Other: Obturator nerve block with ropivacaine 0.2%.
- Obturator nerve block with isotonic salin (Sham Comparator): The same procedure will be performed and 20 milliliters of isotonic saline will be injected in the interfacial plane between the pectineus and external obturator muscles
  Interventions: Other: Obturator nerve block with isotonic saline

INTERVENTIONS:
Other: Obturator nerve block with ropivacaine 0.2%. — 20 milliliters of ropivacaine 2 mg/mL will be injected in the interfacial plane between the pectineus and external obturator muscles.
  Arms: Obturator nerve block with Ropivacaine
Other: Obturator nerve block with isotonic saline — 20 milliliters of isotonic saline will be injected in the interfacial plane between the pectineus and external obturator muscles.
  Arms: Obturator nerve block with isotonic salin

SUMMARY:
Interest of obturator nerve block for analgesia in total hip arthroplasty remains controversial. This regional anesthesia procedure could provide post-operative pain relief as obturator nerve is responsible for innervation of the internal part of the hip joint capsule.

This randomized double-blind study aims to assess obturator nerve block for post-operative analgesia in total hip arthroplasty.

Before the surgery, an ultrasound guided obturator nerve block will be performed with either 20cc of saline or ropivacaine 0.2% (a long-acting local anesthetics). After regional anesthesia, a general anesthesia will be performed for intraoperative period.

This study aims to assess post-operative pain management during the first 24 hours. Ability to walk the day of the surgery will also be collected.

DETAILED DESCRIPTION:
The best strategy to provide post-operative analgesia in total hip arthroplasty (THA) remains controversial. Many procedures have been descripted.

Recent anatomical studies have reported that obturator nerve provide innervation of the internal part of the hip joint capsule. Obturator nerve block could be of major interest as it might improve post-operative analgesia without providing motor block of the quadriceps muscle. This could be associated with an early ability to walk and enhanced recovery.

This randomized double-blind study aims to assess obturator nerve block after THA.

After information, written informed consent will be obtained from all subjects before inclusion. At patient arrival in the anesthetic room, the research assistant will check the patient's consent. Using a computer-generated random number table, patients will be randomized in two-treatment groups by resource not part of the study.

We have planned to include patients aged ≥18 years who were scheduled for primary THA under general anesthesia at the Elective Surgery Center, Clinique Medipole Garonne, Toulouse, France. The Elective Surgery Center annually performs approximately 1500 total hip arthroplasties.

Exclusion criteria are revision of hip arthroplasty, pregnancy, breast feeding, significant psychiatric disturbances, history of relevant drug allergy, chronic pain, current use oral morphine or equivalents.

Obturator nerve block will be performed before general anesthesia as descripted by Nielsen (RAPM, 2019). A linear transducer (X-Porte, Fujifilm SonoSite, Bothell, Washington, USA) will be oriented in the transverse plane and placed in the inguinal crease. The tail of the transducer will be tilted distal in order to visualize the pectineus muscle (medial to the femoral vessels) at its insertion at the superior pubic ramus superficial to the external obturator muscle. An 80 mm nerve block needle (SonoPlex, PAJUNK Medizintechnologie, Geisingen, Germany) will be inserted in-plane from the lateral end of the transducer and advanced until the tip of the needle will be inside the interfascial plane between the pectineus and the obturator externus muscles. 20 milliliters of either ropivacaine 2 mg/mL or isotonic saline-depending on random group allocation-will be injected in the interfacial plane between the pectineus and external obturator muscles. Medication will be prepared by a staff member who won't be involved in the study and delivered in unidentifiable syringes.

As is common in our practice for patients undergoing THA, a standardized general anesthetic technique will be used for all patients including pre-administration of dexmedetomidine (1µg/kg) over 30 minutes, induction with ketamine (0.5 mg/kg), propofol (~3 mg/kg), and dexamethasone (0.15 mg/kg) and maintenance with continuous propofol (~7 mg/kg).

All patients received a standardized intra-operative analgesic strategy including systemic acetaminophen 1000mg, ketoprofen 100mg and nefopam 20mg. A local infiltration of local anesthetics (ropivacaine 0.2%) will be performed by the surgeon as descripted by Kerr. The first injection will be performed into the tissues around the rim of the acetabulum, focusing on both the joint capsule if it remains, and around the exposed gluteal and adductor muscles. The second injection will be made into the external rotators, gluteus tendon, and iliotibial band. The third injection will be made into the subcutaneous tissues under the wound.

In the post-anesthesia care unit (PACU), patients will be assessed for pain using a verbal rating scale (VRS) (VRS, 0=no pain, 10=worst pain). Patients suffering from pain (VRS > 4/10) will receive oxycodone 2 mg intravenous boluses / 3 minutes.

Postoperative analgesic regimen for the first 24 hours' period will include acetaminophen 1000 mg orally every 6 hours, ibuprofen 400 mg orally every 8 hours and oxycodone 10 mg orally every 6 hours in case of VRS > 4/10.

Pain and adverse effects will be assessed each 6 hours during the first 24 hours. The day of the surgery, the ability to ambulate will be assessed by physiotherapists using a 4 point scale (0: Unable to get up; 1: walk <10m; 2: walk between 10 - 50m; 3: walk > 50m).

Patient's follow up ends at either the 24th hour of hospitalization or at patient discharge in day case surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Primary THA under general anesthesia
* Consent for participation
* Affiliation to the french social security system

Exclusion Criteria:

* Revision of hip arthroplasty
* Significant psychiatric disturbances
* Minor patient
* Pregnancy
* Breastfeeding
* Patient is in exclusion period as determined by previous study
* Contraindication to any drug used in the protocol: acetaminophen, ketoprofen, nefopam, oxycodone, propofol, ketamine, Ropivacaine…
* Chronic pain
* Current use oral morphine or equivalents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Oxycodone requirement in PACU | Length of stay in PACU
  In the PACU, patients will be assessed for pain using a verbal rating scale (VRS) (VRS, 0=no pain, 10=worst pain). Patients suffering from pain (VRS > 4/10) will receive oxycodone 2 mg intravenous boluses / 3 minutes.
  Oxycodone requirement will be compared between interventional and control groups.

SECONDARY OUTCOMES:
Pain assessement | Postoperative period : maximum 24 hours after surgery
  Pain will be assessed every 6 hours using a VRS verbal rating scale ranging from 0 to 10 (0=no pain, 10=worst possible pain)
Postoperative Oxycodone consumption | Postoperative period : maximum 24 hours after surgery
  Oxycodone requirement will be compared between interventional and control groups.
Ability to walk | Postoperative period : maximum 24 hours after surgery
  The day of the surgery, the ability to ambulate will be assessed by physiotherapists using a 4-point scale (0: Unable to get up; 1: walk <10m; 2: walk between 10 - 50m; 3: walk > 50m).
Side effects of opioids | Postoperative period : maximum 24 hours after surgery
  Collect side effects associated with Oxycodone: nausea/vomiting, dizziness, urinary retention

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Medipole Garonne, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marty P, Chassery C, Rontes O, Vuillaume C, Basset B, Merouani M, Marquis C, Delussy A, Delbos MC, Ferre F, Bataille B, Joshi G, Delbos A. Obturator nerve block does not provide analgesic benefits in total hip arthroplasty under multimodal analgesic regimen: a randomized controlled trial. Reg Anesth Pain Med. 2021 Aug;46(8):657-662. doi: 10.1136/rapm-2021-102531. Epub 2021 May 5. PMID 33952684